CLINICAL TRIAL: NCT04758312
Title: A Mobile Intervention Merging Yoga and Self-Management Skills (MY-Skills Mobile) for Older Adults With Multiple Chronic Conditions and Their Care-Partners
Brief Title: A Mobile Intervention Merging Yoga and Self-Management Skills
Acronym: MYSkillsMobile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado State University (Other); Clemson University (Other); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-2632
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MY-Skills Mobile Intervention (Experimental): MY-Skills Mobile is an 8-week intervention merging yoga and self-management offered via remote tools including Zoom (video-conferencing software), Canvas (education software), and Qualtrics (survey software) that can be accessed via a computer or tablet. The self-management content is delivered primarily through asynchronous tools that include educational videos and interactive activities for goal setting, action plan, monitoring goals, and problem-solving practice. Yoga is offered synchronously via Zoom two-times per week for 60 minutes (120 minutes per week). The synchronous yoga sessions will be offered at a time that best accommodates participants' schedules. Yoga will become progressively challenging over the eight weeks and will include seated and standing postures.
  Interventions: Behavioral: MY-Skills Mobile

INTERVENTIONS:
Behavioral: MY-Skills Mobile — Yoga and Self-Management Education

SUMMARY:
Chronic disease self-management interventions and meditative movement approaches (.e.g., yoga) can independently improve depressive symptoms. However, to our knowledge there are no interventions integrating evidence-based chronic disease management strategies with yoga to maximize physical, psychological or social outcomes, nor are mobile health platforms commonly used to improve the reach of these integrated interventions. Therefore, we developed Merging-Yoga for Self-Management Skills Mobile (MY-Skills Mobile). Our first aim is to adapt the MY-Skills Mobile to tailor the intervention to older adults with multiple chronic conditions (MCC) by convening a panel of patient and care-partner stakeholders. We will convene four patient and care-partner dyads (N=8) to serve as study partners for three longitudinal focus groups to suggest and review MY-Skills Mobile adaptations. We will then conduct a usability study of MY-Skills Mobile with older adults with MCC and their care-partners. We will conduct two waves of rapid-cycle prototyping with 5 dyads in each wave (N=20). Dyads will participate in MY-Skills Mobile modules. We will then use acceptability surveys and use data in each wave to iteratively adapt MY-Skills Mobile to optimize usability and acceptability.

ELIGIBILITY:
Older Adults with Multiple Chronic Conditions (MCC) and Depressive Symptoms:

* over the age of 65 at time of recruitment
* Multiple chronic conditions: Bayliss Disease Burden/Morbidity Assessment by Self-Report diagnosis > 2 and a disease burden score >2 indicating the presence of at least two chronic conditions that limit activities of daily of living.
* Presence of depressive symptoms will be screened by the Patient Health Questionnaire-2 Scale (PHQ-2), with a score of > 3 indicating at least mild depressive symptoms.
* Participants must be community dwelling
* Live in the United States
* Speak English
* Participants must be able to provide informed consent and have the ability to stand with or without an assistive device.
* We will also use the Patient Activity Readiness Questionnaire (PAR-Q) to determine the safety or possible risk of participation.

Care-Partners:

* Care-partners include any family, friend, or social support that the older adult identifies
* at least age 18
* Can provide informed consent
* Participants must be able to provide informed consent and have the ability to stand with or without an assistive device.
* We will also use the Patient Activity Readiness Questionnaire (PAR-Q) to determine the safety or possible risk of participation.

Exclusion Criteria for Older Adults with MCC and Care-Partners:

* Self-reported diagnosis of Alzheimer's disease or dementia
* Self-reported diagnosis of a severe mental health problem (e.g. schizophrenia, bipolar affective disorder or other psychotic illness)
* Consistent yoga >120 minutes a week
* Completed self-management education in the last year

Participants will not be excluded due to limited technology access. We will provide temporary tablets and mobile hotspot connectivity to interested participants that do not have hardware or internet access.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
User Mobile Application Rating Scale | 8 Weeks
  Usability; 20 items; Range 0-25, Higher score indicates better usability

SECONDARY OUTCOMES:
Patient Health Questionaire-8 | 8 weeks
  Depressive Symptoms; 8 items; Range 0-24; Higher score indicates worse depression
PROMIS Physical Function | 8 weeks
  Physical Function; 20 items with 4 additional global items; Range 0-120; Higher scores indicate better function
PROMIS Self-Efficacy for Managing Chronic Conditions | 8 weeks
  Self-Efficacy; 24 items; Range 0-120; Higher scores indicate better self-efficacy
PROMIS Companionship, Emotional, Instrumental Support | 8 weeks
  Social Support; 14 items, Range 0-70; Higher scores indicate better social support

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Portz, PhD, MSW, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided